CLINICAL TRIAL: NCT00884858
Title: Use of Maraviroc (MVC) in Immunological Non-responder HIV-1-infected Patients.
Brief Title: Maraviroc in Immunological Non-Responder (INR) HIV-1-infected Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ASST Fatebenefratelli Sacco (Other)
Responsible Party: Principal Investigator, Stefano Rusconi, Researcher/Aggregate professor in infectious diseases, ASST Fatebenefratelli Sacco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLS/MVC01/2008
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: HIV Infections
Keywords: HIV-1; CD4; INR; HIV-1 infection; extreme immunological compromission; treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Maraviroc (Experimental): Subjects in this group will add Maraviroc to their current HAART.
  Interventions: Drug: Maraviroc
- 2 (No Intervention): Subjects in this group will continue their current HAART without adding Maraviroc.

INTERVENTIONS:
Drug: Maraviroc — Maraviroc is administered BID according to the other drugs within HAART; dosage ranges from 150 mg to 600 mg bid.
  Other Names: Maraviroc brand name in the EC is Celsentri.
  Arms: Maraviroc

SUMMARY:
Suboptimal improvement in cluster of differentiation 4 (CD4) cell count is not uncommon in HIV-1-infected patients with suppressed plasma HIV-Ribonucleic acid (RNA) levels, and a decrease in CD4 cell count in patients with suppressed or low level viremia has been observed.

Although the efficacy of current antiretroviral medications is well established, some antiviral combinations are very effective in suppressing HIV-1 load whereas do not exert any effect on immune reconstitution.

Both T-cell immune activation and fibrosis of peripheral lymphoid tissue could create an environment in which CD4 T cell count decrease in the setting of low or suppressed plasma viremia is likely to occur.

Another fascinating hypothesis, which has still to be elucidated, is that reconstitution of the depleted CD4 pool is blocked by an excess of glycoprotein 120 (gp120) HIV-1 protein. This extra-production could be counteracted by an inhibitor of the chemokine (C-C motif) receptor 5 (CCR5) co-receptor that represents one of the major docking tools of HIV-1.

With this in mind, the investigators would like to propose and design a pilot exploratory clinical trial involving a population of HIV-1-infected patients that rapidly reached a virologic suppression without a reconstitution of their immune system.

DETAILED DESCRIPTION:
Objectives:

* Evaluate the clinical efficacy of HAART intensification with MVC as treatment of HIV-1 infection in patients with a CD4 count ≤ 200 cells/uL and/or a recovery of CD4 cells < 25% compared to the HAART initiation and with a complete and stable virologic suppression after 12 months of HAART. Patients could also being included if their CD4 slope has been stable without any improvement, with an absolute value around 200 cells/uL.
* Evaluate the effects of HAART intensification with MVC on the modification of immunologic and virologic parameters.
* Evaluate the tolerability of HAART intensification with MVC and the appearance of drug-related side effects.

Design:

This will be a randomised, multicenter, study that will evaluate HAART intensification with MVC as treatment of HIV-1 infection in patients with a CD4 count ≤ 200 cells/uL and/or a recovery of CD4 cells < 25% compared to the HAART initiation and/or a stable CD4 slope without any improvement, with an absolute value around 200 cells/uL and with a complete and stable virologic suppression after 12 months of HAART.

ELIGIBILITY:
Inclusion Criteria:

* age > or = 18
* HIV-Abs positivity detected by ELISA and confirmed by Western-Blot
* CD4 lymphocytes < 200/uL and/or CD4 recovery < 25% after at least 12 months of stable HAART
* HIV-RNA < 50 cp/mL during the last 12 months
* negative pregnancy test at least 14 days prior to treatment
* understanding and signing the informed consent

Exclusion Criteria:

* allergy/intolerance to the study drug
* less than 1 year from any treatment with immunomodulatory agents
* current OIs or neoplasms
* current CVD or EKG abnormalities
* current respiratory tract diseases or COPD
* treatment with steroids within 4 weeks from treatment beginning
* suspect of autoimmune disorder or chronic inflammatory disease
* active IVDUs or alcohol addicts
* AST and ALT > 2.5 ULD
* serum creatinine > 1.5 ULD
* ANC < 1000/uL
* hemoglobin < 10 g/dL
* platelets < 75.000/uL
* reticulocytes > 2%
* Karnofsky score < 50

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
CD4 counts > 200/uL or recovery of CD4 > 25% in 2 consecutive time-points. | 3 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Rusconi, M.D., Principal Investigator — Universita' degli Studi di Milano, Italy
Locations (20):
- Italy (20):
  - Servizio Regionale di Immunologia Clinica e Tipizzazione Tissutale, Azienda Ospedaliero-Universitaria, Torrette Di Ancona, AN
  - Clinica di Malattie Infettive, Policlinico, Universita' degli Studi, Bari, BA
  - Clinica di Malattie Infettive e Tropicali, Università degli Studi di Brescia, Spedali civili, Brescia, BS
  - Divisione di Malattie Infettive, Ospedale S. Maria Annunziata, Antella, FI
  - Clinica di Malattie Infettive, Ospedale San Martino, Genova, GE
  - Divisione di Malattie Infettive, Ospedale San Gerardo, Monza, MB
  - Polo di Medicina Chirurgia e Odontoiatria, Polo Didattico S. Paolo, Milan, MI
  - U.O di Malattie Infettive, Fondazione San Raffaele del Monte Tabor, Milan, MI
  - Divisione Clinicizzata di Malatie Infettive, Azienda Ospedaliera-Polo Universitario "Luigi Sacco", Milan, MI
  - I e II Divisione Malattie Infettive, Azienda Ospedaliera-Polo Universitario Luigi Sacco, Milan, MI
  - Clinica delle Malattie Infettive, Policlinico Universitario, Modena, MO
  - Divisione Dipartimento Urgenze Infettivologiche ad Alta Complessità e correlate all'AIDS, Ospedale Cotugno, Napoli, Napoli
  - U.O. Malattie Infettive, Ospedale S. Spirito, Pescara, PE
  - Clinica delle Malattie Infettive, Policlinico Monteluce, Perugia, PG
  - Clinica delle Malattie Infettive, Policlinico "Tor Vergata", Roma, RM
  - III Divisione di Malattie Infettive, I.N.M.I Lazzaro Spallanzani, Roma, RM
  - IV Divisione di Malattie Infettive, INMI Lazzaro Spallanzani, Roma, RM
  - U.O. Malattie Infettive, Azienda Policlinico Umberto I, Roma, RM
  - Istituto Clinica delle Malattie Infettive, Università Cattolica del Sacro Cuore, Roma, RM
  - Clinica delle Malattie Infettive ,Ospedale Amedeo di Savoia, Torino, TO

REFERENCES:
- [Derived] Rusconi S, Vitiello P, Adorni F, Colella E, Foca E, Capetti A, Meraviglia P, Abeli C, Bonora S, D'Annunzio M, Di Biagio A, Di Pietro M, Butini L, Orofino G, Colafigli M, d'Ettorre G, Francisci D, Parruti G, Soria A, Buonomini AR, Tommasi C, Mosti S, Bai F, Di Nardo Stuppino S, Morosi M, Montano M, Tau P, Merlini E, Marchetti G. Maraviroc as intensification strategy in HIV-1 positive patients with deficient immunological response: an Italian randomized clinical trial. PLoS One. 2013 Nov 14;8(11):e80157. doi: 10.1371/journal.pone.0080157. eCollection 2013. PMID 24244635